CLINICAL TRIAL: NCT06350643
Title: The Quit and Screen Project
Brief Title: Quit and Screen Project
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Virginia Commonwealth University (Other); Coalition for a Tobacco Free Arkansas (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Medical Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 287064; P50MD017319-03S1 (NIH)
Record Dates: First submitted 2024-03-06; First posted 2024-04-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Knowledge; Attitudes; Behavioral Intention
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quit and Screen Project training alone (Experimental): Providers in this arm will only complete the Quit and Screen Project training. This online course will be developed for healthcare providers and will fill gaps in knowledge and attitudes toward lung cancer screening and smoking not covered by the G02 (Global Knowledge Center for Lung Cancer) Lung Cancer Screening training .
  Interventions: Other: Quit and Screen Project training
- Quit and Screen Project training + G02 Lung Cancer Screening training (Experimental): In this arm, providers will complete the G02 (Global Knowledge Center for Lung Cancer) Lung Cancer Screening training and the Quit and Screen Project training. The Quit and Screen Project training is an online course being developed to fill gaps in knowledge and attitudes toward lung cancer screening and smoking not covered by the G02 Lung Cancer Screening training.
  Interventions: Other: Quit and Screen Project training; Other: G02 (Global Knowledge Center for Lung Cancer) Lung Cancer Screening training

INTERVENTIONS:
Other: Quit and Screen Project training — This online course will be developed for healthcare providers and will fill gaps in knowledge and attitudes toward lung cancer screening and smoking not covered by the G02 (Global Knowledge Center for Lung Cancer) Lung Cancer Screening training.
Other: G02 (Global Knowledge Center for Lung Cancer) Lung Cancer Screening training — The G02 (Global Knowledge Center for Lung Cancer) Lung Cancer Screening training is an online course that covers disparities in lung cancer and smoking, patient barriers to lung cancer screening, and provider resources for addressing common barriers.
  Arms: Quit and Screen Project training + G02 Lung Cancer Screening training

SUMMARY:
The Quit and Screen Project seeks to engage healthcare providers in helping adults who smoke to quit tobacco use, including menthol cigarettes and flavored cigars, and screen for lung cancer early as strategies to reduce multiple chronic diseases.

The goal of this clinical trial is to test the feasibility and impact of the Quit and Screen Project alone versus the G02 (Global Knowledge Center for Lung Cancer) Lung Cancer Screening training + the Quit and Screen Project training modules on changes in provider knowledge, attitudes, and behavioral intentions related to provider advice to quit smoking and referrals for low dose computed tomography among health care providers randomly assigned to each condition. Participants will complete the training modules and complete pre- and post-tests to assess these outcomes.

DETAILED DESCRIPTION:
This clinical trial tests the feasibility and impact of the Quit and Screen Project alone versus the G02 (Global Knowledge Center for Lung Cancer) Lung Cancer Screening training + the Quit and Screen Project training modules on changes in provider knowledge, attitudes, and behavioral intentions related to provider advice to quit smoking and referrals for low dose computed tomography among health care providers randomly assigned to each condition.

In partnership with the National Medical Association, investigators will recruit 300 healthcare providers who provide clinical services to individuals who smoke smoke. Interested providers will be screened; if eligible, the will complete informed consent. Providers who complete the online consent and agree to enroll in the training study will be individually randomized to one of 2 conditions: The Quit and Screen Project alone versus the G02 (Global Knowledge Center for Lung Cancer) Lung Cancer Screening training + the Quit and Screen Project training. After randomization, providers will complete a pre-test assessing their knowledge, attitudes, and behavioral intentions related to provider advice to quit smoking and referrals for low dose computed tomography. Providers will then complete an online training. Providers will then complete a post-test assessing their 1) knowledge, attitudes, and behavioral intentions related to provider advice to quit smoking and referrals for low dose computed tomography and 2) preferences for the online materials and satisfaction with the training. Feasibility will be assessed using data on provider interest in the training and training reach.

ELIGIBILITY:
Inclusion Criteria:

* Current National Medical Association (NMA) member
* Serves a patient clientele who smokes
* At least 20% of time (1 day per week) devoted to clinical care
* Currently screens clients for tobacco use in the clinic
* Have the capacity to refer smokers to a patient navigator
* Willing to provide informed consent
* Will provide contact email, address and phone.

Exclusion Criteria:

* None

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Familiarity with treatment guidelines for tobacco and nicotine treatment | This is pre-post design where participants will complete a pre-test immediately before completing a 30-60 minute online training and then a post-test immediately after completing training.
  Familiarity with treatment guidelines was assessed using an modified question from the Healthcare Provider Survey published by Primary Care Development Corporation in 2008.
Weaver et al. 2012 Provider Attitudes and Perceptions about smoking cessation | This is pre-post design where participants will complete a pre-test immediately before completing a 30-60 minute online training and then a post-test immediately after completing training.
  These questions assessed providers perceptions about the benefits of smoking cessation and the benefits of providers advising patients to quit smoking.
Weaver et al. 2012 Provider Perceptions about provider barriers to providing smoking cessation interventions to patients | This is pre-post design where participants will complete a pre-test immediately before completing a 30-60 minute online training and then a post-test immediately after completing training.
  Perceptions about provider barriers to addressing smoking cessation with patient were assessed using modified questions from a questions published in Weaver et al. 2012, Carter-Harris et al. (2017), and Raz et al. 2019.
Provider Perceptions about patient barriers to smoking cessation | This is pre-post design where participants will complete a pre-test immediately before completing a 30-60 minute online training and then a post-test immediately after completing training.
  Perceptions about patient barriers to smoking cessation were assessed using modified questions from a questions published in Weaver et al. 2012, Carter-Harris et al. (2017), and Raz et al. 2019.
Behavioral intentions to screen and advise patients about smoking cessation | This is pre-post design where participants will complete a pre-test immediately before completing a 30-60 minute online training and then a post-test immediately after completing training.
  A set of questions based on the Theory of Planned Behavior assessed provider's intention to screen patients for tobacco use and provide them interventions and referrals for treatment.
Familiarity with lung cancer screening guidelines | This is pre-post design where participants will complete a pre-test immediately before completing a 30-60 minute online training and then a post-test immediately after completing training.
  Familiarity with treatment guidelines was assessed using an modified question from the Healthcare Provider Survey published by Primary Care Development Corporation in 2008.
Knowledge about low dose computed tomography for lung cancer screening | This is pre-post design where participants will complete a pre-test immediately before completing a 30-60 minute online training and then a post-test immediately after completing training.
  Familiarity with treatment guidelines was assessed using an modified question from the questions published by Kota et al. 2022, Carter-Bawa et al. 2022, and the National Cancer Institute National Survey of Primary Care Physicians' Recommendations & Practices for Breast, Cervical, Lung, & Colorectal Cancer Screening.
Perceptions about shared decision-making for low dose computed tomography for lung cancer screening | This is pre-post design where participants will complete a pre-test immediately before completing a 30-60 minute online training and then a post-test immediately after completing training.
  Questions were modified from the questions published by Forcino et al. in 2018.
Perceptions about provider barriers to referring patients to low dose computed tomography for lung cancer screening | This is pre-post design where participants will complete a pre-test immediately before completing a 30-60 minute online training and then a post-test immediately after completing training.
  Questions were modified from questions published by Coughlin et al. 2020.
Provider Perceptions about patient barriers to get screened for lung cancer | This is pre-post design where participants will complete a pre-test immediately before completing a 30-60 minute online training and then a post-test immediately after completing training.
  Perceptions about patient barriers to getting screened for lung cancer were assessed using modified questions from a questions published in Weaver et al. 2012, Carter-Harris et al. (2017), and Raz et al. 2019.
Behavioral intentions to advise patients to get screened for lung cancer via low dose computed tomography | This is pre-post design where participants will complete a pre-test immediately before completing a 30-60 minute online training and then a post-test immediately after completing training.
  A set of questions based on the Theory of Planned Behavior assessed provider's intention to advise patients who smoke to get screened for lung cancer via low dose computed tomography.

SECONDARY OUTCOMES:
Characteristics of enrolled healthcare providers | This is pre-post design. This outcome will be measured during the pre-test immediately before participants complete the 30-60 minute online training.
  Study process tracking metrics will be used to assess the demographic, training, and clinical practice characteristics of providers who enroll in the training.
Retention: Percent of providers complete the training after enrolling | This is pre-post design where participants will complete a pre-test immediately before completing a 30-60 minute online training and then a post-test immediately after completing training.
  Study process tracking metrics will be used to assess retention of providers who enroll in the training.
Adherence to completing training modules: Percent of modules completed | This is pre-post design where participants will complete a pre-test immediately before completing a 30-60 minute online training and then a post-test immediately after completing training.
  Study process tracking metrics and training completion data will be used to assess the percent of training modules completed (i.e., the number of modules completed divided by the total available modules).
Preferences regarding training | This is pre-post design. This outcome will be measured during the post-test immediately after they complete the 30-60 minute online training.
  Questions will assess provider feedback on the online training module.
Satisfaction with training | This is pre-post design. This outcome will be measured during the post-test immediately after they complete the 30-60 minute online training.
  Questions will assess provider satisfaction on the online training module.

CONTACTS AND LOCATIONS:
Overall Officials: Pebbles Fagan, PhD, MPH, Principal Investigator — University of Arkansas; Mignonne Guy, PhD, Principal Investigator — Virginia Commonwealth University; Ashley Clawson, PhD, Principal Investigator — University of Arkansas
Locations (1):
- Virginia Commonwealth Univesity, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No